CLINICAL TRIAL: NCT06807359
Title: Open-label Clinical Phase 1/2 Study to Assess the Safety and Efficacy of the SpectraCure P18 System and Verteporfin for Injection for the Treatment of Primary Localized Prostate Cancer
Brief Title: Photodynamic Therapy of Primary Localized Prostate Cancer With the SpectraCure P18 System
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SpectraCure AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPC11-02-110
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Photochemotherapy; Verteporfin

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, non-randomized multicenter study without control group.
  Phase 1 - Dose-escalation
  Phase 2 - Cohort expansion
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- PDT with VFI (Experimental): Interstitial Photodynamic Therapy (PDT) and Verteporfin for Injection (VFI)
  Interventions: Device: Photodynamic Therapy (PDT); Drug: Verteporfin Injection

INTERVENTIONS:
Device: Photodynamic Therapy (PDT) — The PDT treatment is provided with the SpectraCure P18 laser light delivery system.
  PDT will be performed during general anesthesia. Optical fibers will be inserted into the prostate with a transperineal approach using transrectal ultrasound guidance. The intent is to deliver an adequate light dose throughout the prostate. Subjects will receive VFI intravenously, approximately 60-90 minutes prior to light delivery. The photosensitizer is activated with light of a specific wavelength that is delivered to the tumor via optical fibers. The activated photosensitizer reacts with oxygen to form highly toxic radicals which induce cell death in the tumour.
  * Phase 1: Light dose escalation. Three subjects will be treated per dose level (20 - 40 J/cm2). If no dose-limiting toxicities occur, dose will be escalated (20 - 40 J/cm2) until the Recommended Phase 2 Dose (RPD2) is established.
  * Phase 2: Cohort expansion with the RPD2.
Drug: Verteporfin Injection — Verteporfin for Injection (VFI), photosensitizing drug, will be administered intravenously at a dose of 15 mg/m2 body surface area.
  Other Names: Visudyne

SUMMARY:
The goal of this study is to obtain safety data, establish dose parameters, and effectiveness of treatment for the SpectraCure P18 System with IDOSE®, together with verteporfin for injection (VFI) as photosensitizer, for the treatment of primary localized prostate cancer.

The study will be divided into two parts, with Phase I, dose-escalation, to study safety and establish an effective light dose, followed by Phase II, cohort expansion, to evaluate clinical efficacy and confirm safety/tolerability. The subjects will be followed for a period of 18 months to determine the primary outcome. The long-term follow-up is an additional 18 months, i.e. a total of 36 months.

Interstitial Photodynamic Therapy (PDT) will be performed during general anesthesia. Optical fibers will be inserted into the prostate with a transperineal approach using transrectal ultrasound guidance. The intent is to deliver an adequate light dose throughout the prostate. Subjects will receive VFI intravenously, approximately 60-90 minutes prior to light delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years.
2. Histologically confirmed organ-confined adenocarcinoma of the prostate cancer diagnosed within the last 9 months. Including subjects on active surveillance with evidence of disease progression and a prostate biopsy not older than 9 months.

   a. This prostate biopsy should be targeted and systematic (transperineal or transrectal are both acceptable) and include both systematic sampling with a minimum of 8 cores (4 right, 4 left) as well as MRI fusion targeted cores. The minimum number of targeted cores is two (2) but more may be included at the discretion of the surgeon.
3. Gleason Score 7 (3+4 or 4+3).
4. PSA ≤ 15 ng/mL.
5. Lesion volume on mpMRI < 1.5 cm3.
6. Adequate stage imaging such as pelvic CT/MRI/PET scan within the last 6 months confirming localized cancer.

   - Bone scan is optional if PSA < 10 ng/mL.
7. Treatment target volume <50 cm3 defined by TRUS or MRI.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Expected survival ≥ 36 months.
10. Sufficient bone marrow reserve as indicated by; granulocyte count ≥ 1500/mm3, platelet count ≥ 100,000/mm3.
11. Adequate renal function as defined by creatinine ≤ 1.5 mg /dl.
12. Adequate hepatic function, based on a total bilirubin ≤ 1.5 mg/dl, serum glutamate-oxaloacetate transaminase (SGOT) ≤ 3 times the upper limit of normal, and alanine transaminase (ALT) ≤ 3 times the upper limit of normal.
13. Signed Informed Consent.

Exclusion Criteria:

1. Evidence of locally advanced, regional pelvic lymph node metastasis, or metastatic disease.
2. Any suspicious for, probable, or definite extracapsular extension on pretreatment MRI
3. Contralateral PIRADS 4/5 lesion (even if negative targeted biopsy)
4. High volume GG1 disease in the contralateral prostate, outside of the ablation zone. High volume is defined as >1 core of GG1 with a linear amount of carcinoma >6mm.
5. Prior radical surgery for carcinoma of the prostate, prior pelvic radiation, prior TURP, prior cryosurgery of the prostate.
6. Prior treatment with any form of brachytherapy.
7. Previous androgen deprivation therapy (ADT) or chemotherapy for prostate cancer.
8. Prior or current bleeding diathesis.
9. Tumors known to be eroding into a major blood vessel in or adjacent to the illumination site.
10. Use of Alpha-reductase inhibitors (ARIs) within 90 days of enrolment.
11. Any serious active or co-morbid medical conditions, laboratory abnormality, psychiatric illness, active or uncontrolled infections, or serious illnesses or medical conditions that would prevent the patient from participating or to be managed according to the protocol (according to investigator's decision).
12. Mental incapacity or psychiatric illness that would interfere with the subject's ability to understand and give informed consent or to complete follow-up visits according to the judgement of the investigator.
13. Contraindication for photosensitizer including:

    1. Porphyria or other diseases exacerbated by light.
    2. Known hypersensitivity to verteporfin for injection (VFI) or to any of the excipients.
    3. Known allergies to porphyrins.
14. On-going therapy with a photosensitizing agent.
15. Enrolment in another therapeutic clinical study within 3 month prior to enrolment and throughout the study.
16. Contraindication for MRI/Gadolinium contrast such as: implants, hip prosthesis, severe renal impairment (glomerular filtration rate [GFR] <30 mL/min/1.73m2), or previous contrast reactions.
17. Has known hypersensitivity to pancuronium bromide, atricurium or cisatricurium

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with primary localized prostate cancer
Enrollment: 43 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment | Within 4 weeks of treatment in each cohort.
  Number of participants with treatment related adverse events as assessed by CTCAE v5.0 related to therapy per protocol.
  Dose limiting toxicities are defined as grade 3 non-hematologic or grade 4 hematologic toxicities that are possibly, probably or definitely related to PDT.
Safety - Damage to the periprostatic tissue mediated by PDT | 5-9 days following PDT
  Potential damage to the periprostatic tissue will be evaluated by contrast-enhanced and not-contrast enhanced MRI.
Treatment efficacy | 6 and 18 months post PDT
  Percentage of subjects with negative in-field biopsies (histopathologically tumor-free)

SECONDARY OUTCOMES:
Adequacy of effectiveness | Within 1 week following PDT
  Extent of quantifiable treatment effect in the prostate evaluated by MRI to determine the extent of necrosis in the prostate
Treatment efficacy | 6 and 18 months post PDT
  Rate of negative in-field biopsy as defined by the Delphi consensus criterion (≤ 3 mm of Gleason ≤ 6 disease in any biopsy core is insignificant).
Device performance | Day of PDT
  Light dose coverage >90% of the target volume; evaluated by dose-volume histograms in >80% of subjects
Percentage of subjects with biochemical failure | 6 and 10 weeks, 6, 18, 24 and 36 months post PDT
  Failure defined as a rise in PSA level of 2.0 ng/mL or more, over and above the nadir
Percentage of subjects with extra prostatic or distant disease | 6 and 18 months post PDT
  Remaining localized tumour will be evaluated by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fainberg, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center, New York, United States
Locations (2):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Klinik für Urologie Universitätsklinikum Köln, Cologne, Germany